CLINICAL TRIAL: NCT02375672
Title: A Multi-Center, Single Arm, Phase II Study of Pembrolizumab (MK-3475) in Combination With Chemotherapy for Patients With Advanced Colorectal Cancer: HCRN GI14-186
Brief Title: Study of Pembrolizumab in Combination With Chemotherapy for Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kathy Miller, MD, Principal Investigator, Hoosier Cancer Research Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GI14-186
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Results first posted 2021-10-08 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Cancer
Keywords: Pembrolizumab; MK-3475
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab (MK-3475) + mFOLFOX6 (Experimental): Following the safety run-in cohort:
  mFOLFOX6 Treatment D1 and D15 (every 2 weeks); Pembrolizumab (MK-3475) IV over 30 minutes (every 3 weeks)
  Interventions: Drug: Pembrolizumab; Drug: mFOLFOX6

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (MK-3475) 200mg IV over 30 minutes every 3 weeks
  Other Names: MK-3475
Drug: mFOLFOX6 — mFOLFOX6 Treatment D1 and D15 (Cycle = 28 days)
  * Oxaliplatin 85 mg/m^2 IV with
  * Leucovorin 400 mg/m^2 IV followed by
  * 5FU 400 mg/m^2 bolus and then 2400 mg/m^2 via continuous infusion

SUMMARY:
This is a multi-institutional, single arm, open-label, phase II study, including a safety run-in cohort. No randomization or blinding involved.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

INVESTIGATIONAL TREATMENT:

mFOLFOX6 Treatment D1 and D15 (Cycle = 28 days)

* Oxaliplatin 85 mg/m2 IV with
* Leucovorin 400 mg/m2 IV followed by
* 5FU 400 mg/m2 bolus and then 2400 mg/m2 via continuous infusion

Pembrolizumab (MK-3475) IV over 30 minutes every 3 weeks

SAFETY RUN-IN COHORT:

The safety run-in cohort will include 6 subjects treated with 200 mg (fixed) IV infusion of pembrolizumab (MK-3475) every 3 weeks plus standard-dose mFOLFOX6 given every 2 weeks. These first 6 subjects will be followed for 4 weeks for dose limiting toxicities (DLT) before enrolling an additional 24 patients. If a DLT is observed in no more than 1 of 6 subjects, the trial will continue with enrolling subjects to the remainder of the phase II portion of the study. Otherwise, 6 additional subjects will be enrolled at dose level -1. If no more than one DLT is observed, then phase II will enroll subjects at dose level -1 for the total expected number of accrual.

Disease evaluation every 8 weeks or after every 2 cycles

Demonstrate adequate organ function as defined by the following laboratory values at study entry. All screening labs should be performed within 14 days prior to registration for protocol therapy.

Hematopoietic:

* Hemoglobin ≥ 9 g/dL (transfusions are acceptable)
* Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
* Platelets ≥ 100 × 10^9/L

Renal:

* Serum creatinine ≤ 1.5 × upper limit of normal (ULN), or measured or calculated creatinine clearance (estimated by Cockcroft-Gault formula below or measured) ≥ 50 mL/min

Hepatic:

* Serum total bilirubin ≤ 1.5 × ULN
* Aspartate aminotransferase (AST, SGOT) and alanine aminotransferase (ALT, SGPT) ≤ 3 × ULN, unless evidence of liver metastases, then AST/ALT ≤ 5 x ULN

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Be ≥ 18 years of age on day of signing informed consent.
* Have a performance status of 0 or 1 on the ECOG Performance Scale within 14 days prior to registration.
* Have histological or cytological evidence of colorectal adenocarcinoma with confirmation of metastatic disease either by pathologic or radiologic findings.
* Have identified tissue from an archival tissue sample (preferably from a metastasis, but sample from primary tumor allowable) or newly obtained core or excisional biopsy of a tumor lesion.
* Have had no prior systemic therapy for advanced or metastatic disease. Prior adjuvant therapy should have been completed at least 9 months from documentation of metastatic disease. Prior palliative radiotherapy allowed if toxicities resolved to grade 1 or baseline.
* Have measurable disease according to RECIST v1.1 obtained by imaging within 28 days prior to registration.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 14 days prior to study registration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Subjects of childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) are those who meet the following criteria: has not undergone a hysterectomy or bilateral oophorectomy; OR has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication

Exclusion Criteria:

* Has clearly resectable colon cancer liver metastases (CCLM), for example oligometastatic disease involving only one lobe of the liver. Subjects with suspected resectable CCLM should undergo evaluation by a liver surgeon prior to enrollment to document the incurable nature of their disease.
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of registration. Subjects are not permitted to participate in another investigational drug study while being treated on this protocol.
* Is unable to receive a port or peripherally inserted central catheter (PICC).
* Has a diagnosis of immunodeficiency or is receiving chronic steroid therapy of prednisone ≥ 10 mg daily or any equivalent dose of corticosteroids.
* Has previously undergone organ or bone marrow transplantation and is on immunosuppressive therapy
* Has had major surgery or significant traumatic injury within 4 weeks of study registration. Subjects must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. A diagnostic or research biopsy does not exclude subjects from enrollment. Placement of a vascular access device such as a Port-A-Cath is not considered major surgery
* Has baseline peripheral neuropathy/paresthesia grade ≥ 1.
* Has a known additional malignancy within the past 3 years. Exceptions include treated localized basal cell or squamous cell carcinoma of the skin, in situ cervical or vulvar carcinoma that has undergone potentially curative therapy, superficial bladder tumors (Ta, Tis & T1), ductal carcinoma in situ (DCIS) of the breast and low grade prostate cancer (Gleason sore 6). Any cancer curatively treated > 3 years prior to registration with no clinical evidence of recurrence is permitted
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to trial registration and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial registration.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions to the rule: subjects with vitiligo; subjects with resolved childhood asthma/atopy; subjects that require intermittent use of bronchodilators or local steroid injections; subjects with hypothyroidism stable on hormone replacement or patients with Sjögren's syndrome
* Has a history of pneumonitis that required steroids or current pneumonitis.
* Has known history of active tuberculosis.
* Has an active infection requiring systemic therapy (≥ grade 2) for more than 3 days within 1 week of enrollment.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of pembrolizumab (MK-3475).
* Has known hypersensitivity to fluorouracil (5FU), oxaliplatin, or other platinum agents.
* Known hypersensitivity to pembrolizumab or any of its excipients.
* Has known dihydropyrimidine dehydrogenase deficiency (DPD) deficiency (testing not required)
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Has known active Hepatitis B unless subject has been on antiviral agents for at least 2 months (baseline testing not required)
* Has a known history of Human Immunodeficiency Virus (HIV) or Hepatitis C (baseline testing is not required).
* Has received a live vaccine within 30 days prior to trial registration.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the site investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has any other psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule. Those conditions should be discussed with the subject before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Safi Shahda, M.D., Study Chair — Hoosier Cancer Research Network
Locations (3):
- United States (3):
  - Emory University: Winship Cancer Institute, Atlanta, Georgia
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab (MK-3475) + mFOLFOX6: Following the safety run-in cohort:
  mFOLFOX6 Treatment D1 and D15 (every 2 weeks); Pembrolizumab (MK-3475) IV over 30 minutes (every 3 weeks)
  Pembrolizumab: Pembrolizumab (MK-3475) 200mg IV over 30 minutes every 3 weeks
  mFOLFOX6: mFOLFOX6 Treatment D1 and D15 (Cycle = 28 days)
  * Oxaliplatin 85 mg/m^2 IV with
  * Leucovorin 400 mg/m^2 IV followed by
  * 5FU 400 mg/m^2 bolus and then 2400 mg/m^2 via continuous infusion
Period: Overall Study
Arm/Group | Pembrolizumab (MK-3475) + mFOLFOX6
Started | 30
Completed | 10
Not Completed | 20
Not completed — remain on follow up | 20

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab (MK-3475) + mFOLFOX6
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 47.5 [28 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead.
  Participants
    0 | 21
    1 | 9
Stage at Presentation [Count of Participants; unit: Participants] — The TNM system helps describe cancer in great detail. But, for many cancers, the TNM combinations are grouped into five less-detailed stages.
  Stage 0: Abnormal cells are present but have not spread to nearby tissue. Also called carcinoma in situ, or CIS. CIS is not cancer, but it may become cancer.
  Stage I, Stage II, and Stage III: Cancer is present. The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Stage IV: The cancer has spread to distant parts of the body.
  Participants
    I | 1
    II A | 2
    II B | 0
    III A | 0
    III B | 2
    III C | 3
    IV | 22
Sites of Metastasis [Number; unit: participants]
  Liver | 22
  Lung | 7
  Lymph Node | 5
  Bone | 2
  Ileum | 3
  Peritoneum | 3
  Other | 5

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (mPFS)
Description: Determine if pembrolizumab (MK-3475) in combination with chemotherapy improves median progression free survival (mPFS) compared to historical standards.
  Response Criteria - Evaluation of target lesions Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: From time of registration to the time of documented progression per RECIST 1.1 or subject death (estimate 14 months)
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | Pembrolizumab (MK-3475) + mFOLFOX6
Number analyzed (Participants) | 30
months | 8.8 [7.7 to 11.3]

2. Secondary Outcome: Disease Assessment for Objective Response Rate (ORR)
Description: To determine the number of patients who achieve complete response and partial response per irRC criteria.
Time Frame: Begin C1D1 and every 8 weeks thereafter (up to 24 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab (MK-3475) + mFOLFOX6
Number analyzed (Participants) | 30
Participants | 17

3. Secondary Outcome: Disease Assessment for Disease Control Rate
Description: Disease control rate (DCR), defined as the sum of subjects with complete response, partial response and stable disease per RECIST 1.1 criteria.
Time Frame: Begin C1D1 and every 8 weeks thereafter (up to 24 months) per RECIST 1.1 criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab (MK-3475) + mFOLFOX6
Number analyzed (Participants) | 30
Participants | 30

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) reported as number of subject alive at a median followup time of 19.9 months.
Time Frame: Subject should be followed from time of registration till the time of subject death up to a maximum 35.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab (MK-3475) + mFOLFOX6
Number analyzed (Participants) | 30
Participants
  Alive | 20
  Expired | 10

5. Secondary Outcome: Number of Patients With Grade 3 or Higher Treatment Related Adverse Event
Description: To assess safety and tolerability of mFOLFOX6 and pembrolizumab (MK-3475) combination chemotherapy in patients with advanced colorectal cancer per CTCAE v4.0.
  Events are considered related if they assessed possible, probable or definite with study drug.
Time Frame: Begin C1D1 and very 2 weeks (Day 1) for up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab (MK-3475) + mFOLFOX6
Number analyzed (Participants) | 30
Participants | 15

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) was reported from the time of consent and until 30 days after last dose of study drug up to a maximum 108 weeks.
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) v4 were utilized for AE reporting
Arm/Group | Pembrolizumab (MK-3475) + mFOLFOX6
All-Cause Mortality (participants affected / at risk) | 10/30
Serious Adverse Events (participants affected / at risk) | 7/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (MK-3475) + mFOLFOX6 (N=30)
ANAPHYLAXIS (Immune system disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
ENDOCRINE DISORDERS (Endocrine disorders) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 3 (3)
FEVER (General disorders) | 1 (1)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (2)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (MK-3475) + mFOLFOX6 (N=30)
ABDOMINAL PAIN (Gastrointestinal disorders) | 10 (16)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 (13)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 (6)
ALLERGIC REACTION (Immune system disorders) | 1 (1)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3)
ANEMIA (Blood and lymphatic system disorders) | 5 (7)
ANOREXIA (Metabolism and nutrition disorders) | 8 (16)
ANXIETY (Psychiatric disorders) | 2 (2)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7 (12)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4)
BLOATING (Gastrointestinal disorders) | 2 (2)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 6 (11)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
BUTTOCK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
CHILLS (General disorders) | 4 (6)
CONJUNCTIVITIS (Eye disorders) | 1 (2)
CONSTIPATION (Gastrointestinal disorders) | 10 (15)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (8)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 3 (4)
DIARRHEA (Gastrointestinal disorders) | 14 (31)
DRY MOUTH (Gastrointestinal disorders) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
DYSESTHESIA (Nervous system disorders) | 2 (3)
DYSGEUSIA (Nervous system disorders) | 6 (7)
DYSPEPSIA (Gastrointestinal disorders) | 5 (5)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
EDEMA LIMBS (General disorders) | 3 (4)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 1 (1)
EYE DISORDERS (Eye disorders) | 1 (1)
EYE PAIN (Eye disorders) | 1 (1)
FACIAL PAIN (General disorders) | 1 (1)
FATIGUE (General disorders) | 18 (63)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FECAL INCONTINENCE (Gastrointestinal disorders) | 1 (2)
FEVER (General disorders) | 5 (8)
GAIT DISTURBANCE (General disorders) | 1 (1)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 3 (3)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 3 (3)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
HALLUCINATIONS (Psychiatric disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 6 (8)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 8 (35)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 3 (4)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3 (4)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPOTENSION (Vascular disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 3 (4)
INFUSION RELATED REACTION (General disorders) | 2 (3)
INSOMNIA (Psychiatric disorders) | 2 (4)
LIP PAIN (Gastrointestinal disorders) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 3 (11)
MUCOSITIS ORAL (Gastrointestinal disorders) | 10 (15)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 3 (4)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (2)
NAUSEA (Gastrointestinal disorders) | 22 (37)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 6 (15)
NEUTROPHIL COUNT DECREASED (Investigations) | 10 (21)
ORAL PAIN (Gastrointestinal disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 (3)
PAPULOPUSTULAR RASH (Infections and infestations) | 2 (2)
PARESTHESIA (Nervous system disorders) | 4 (4)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 19 (68)
PLATELET COUNT DECREASED (Investigations) | 8 (26)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 3 (4)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 4 (4)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4 (4)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 5 (10)
RECTAL PAIN (Gastrointestinal disorders) | 2 (2)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SINUS PAIN (Nervous system disorders) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 3 (3)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 3 (3)
SYNCOPE (Nervous system disorders) | 1 (1)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
VOMITING (Gastrointestinal disorders) | 9 (13)
WEIGHT GAIN (Investigations) | 2 (2)
WEIGHT LOSS (Investigations) | 5 (5)
WHITE BLOOD CELL DECREASED (Investigations) | 5 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT02375672/Prot_SAP_000.pdf